CLINICAL TRIAL: NCT06726837
Title: Effect of Epoxy Resin-Based and Bioceramic-Based Root Canal Sealers on Postoperative Pain: A Randomized Controlled Clinical Trial
Brief Title: Effect of Different Root Canal Sealers on Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Merve YENICERI OZATA, Associate Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUFD-END-MYO-01; DİŞ.24.013 (Other Grant/Funding Number: Dicle University Scientific Research Projects Coordination)
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Dental Pain; Root Canal Obturation; Warm Vertical Compaction; Root Canal Sealers; Visual Analog Scale
Keywords: Postoperative pain; AH Plus; Bio-C Sealer; TotalFill BC Sealer; visual analog scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will blinded to the group to which they will assigned, but the operator will aware of it. Outcome assessments will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: AH Plus Root Canal Sealer (Active Comparator): Patients will be informed and have an informed consent form signed. Infiltrative anesthesia (4% articaine hydrochloride containing 1:100,000 adrenaline) will be applied. The relevant tooth will be isolated, and the access cavity will be prepared.
  The canal length will be determined, and canals will be prepared with Reciproc R25 files. 15 ml of 2.5% sodium hypochlorite (NaOCl) will be used. In the final irrigation, 5 ml of 17% EDTA, 5 ml of 2.5% NaOCl, and 2 ml of distilled water will be used and activated with a sonic activation device.
  All canals will be filled using the warm vertical condensation technique and AH Plus root canal sealer (n=24). All treatments will be completed in a single session.
  Patients will be given a visual analog scale (VAS) form and asked to mark their pain levels between 0 and 10 at 6, 24, 48, 72 hours, and 7 days after treatment. At the end of the 7th day, patients will be called for a check-up, and VAS questionnaires will be collected.
  Interventions: Other: Postoperative pain - 6th hour; Other: Postoperative pain - 24th hour; Other: Postoperative pain - 48th hour; Other: Postoperative pain - 72nd hour; Other: Postoperative pain - 7 day
- Group 2: TotalFill BC Sealer (Active Comparator): All anesthesia, isolation, root canal preparation procedure, and filling technique are the same as in group 1. However, TotalFill BC root canal sealer will be used in this group instead of Ah Plus, which was used in group 1.
  Interventions: Other: Postoperative pain - 6th hour; Other: Postoperative pain - 24th hour; Other: Postoperative pain - 48th hour; Other: Postoperative pain - 72nd hour; Other: Postoperative pain - 7 day
- Group 3: Bio-C Root Canal Sealer (Active Comparator): All anesthesia, isolation, root canal preparation procedure, and filling technique are the same as in group 1. However, Bio-C root canal sealer will be used in this group instead of Ah Plus, which was used in group 1.
  Interventions: Other: Postoperative pain - 6th hour; Other: Postoperative pain - 24th hour; Other: Postoperative pain - 48th hour; Other: Postoperative pain - 72nd hour; Other: Postoperative pain - 7 day

INTERVENTIONS:
Other: Postoperative pain - 6th hour — Patients will be given the VAS Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 6th hour.
Other: Postoperative pain - 24th hour — Patients will be given the VAS Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 24th hour.
Other: Postoperative pain - 48th hour — Patients will be given the VAS Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 48th hour.
Other: Postoperative pain - 72nd hour — Patients will be given the VAS Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 72nd hour.
Other: Postoperative pain - 7 day — Patients will be given the VAS Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 7 day.

SUMMARY:
This randomized clinical study aims to compare postoperative pain in patients after root canal treatments using different root canal filling materials.The root canal pastes that will be tested for postoperative pain in this study have been used worldwide for many years.

Seventy-two patients with single-rooted teeth without pain symptoms but diagnosed with pulpitis and without any previous fillings or prostheses will be randomly divided into three groups according to the root canal sealers. Then the teeth in these groups will be treated with three different root canal sealers. Endodontic treatment will be performed in a single session, following standardized preparation and irrigation protocols, using the warm vertical condensation technique on all teeth.

Patients will be given a Visual Analog Pain Assessment Scale and asked to mark their pain levels between 0 and 10 at 6, 24, 48, 72 hours, and 7 days after root canal treatment. Patients will be called for a check-up at the end of the 7th day, and VAS questionnaires will be collected.

The investigators will be made to determine which root canal sealer causes the least pain.

The null hypothesis of this study was that there would be no difference in post-procedure pain between the groups.

DETAILED DESCRIPTION:
This study will include 72 participants who apply to the Department of Endodontics, Faculty of Dentistry, Dicle University, with the need for root canal treatment, and who meet the inclusion and exclusion criteria specified. Root canal treatment will be applied only to the single-rooted and single-canal teeth of these patients in the lower jaw. Patients will be informed before the procedure, and an informed consent form will be signed. Block anesthesia (4% articaine hydrochloride containing 1:100,000 adrenaline) will be applied to the lower jaw, the relevant tooth will be isolated with a rubber dam, caries, and existing restorations will be removed with high-speed diamond burs under water cooling, and the access cavity will be prepared. The root canal length will be determined using an apex locator and a size 8 or 10 K-file and confirmed radiographically. Initial root canal shaping will be done with a size 20 K file, followed by a nickel-titanium file system Reciproc R25 in the "RECIPROC ALL" mode with a working length. Additional instrumentation will be done with R40 files according to the initial apical diameter. A total of 15 ml of 2.5% sodium hypochlorite (NaOCl), the worldwide gold standard root canal irrigation solution, will be used with a 30-gauge irrigation needle (TruNatomy, Dentsply Sirona). In all irrigation procedures, the irrigation needle will be placed 2 mm shorter than the canal's working length and applied with moderate pressure to prevent irrigation accidents. Finally, final irrigation will be performed with 5 ml 17% EDTA (a chelator commonly used during root canal treatment), 5 ml 2.5% NaOCl, and 2 ml distilled water, respectively. During the final irrigation process, irrigation activation will be performed for 30 seconds with a sonic irrigation activation device. Finally, the root canals will be dried with paper points. Then, the patients will be randomly divided into three treatment groups according to the root canal sealer used (n=24).

Group 1: AH Plus Root Canal Sealer (Dentsply Sirona, Ballaigues, Switzerland) Group 2: TotalFill BC Sealer (FKG Dentaire, La Chaux-des-Fonds, Switzerland) Group 3: Bio-C Sealer (Angelus, PR, Brazil).

The determined root canal sealer will be sent to the canals. Then, all canals will be filled using the hot vertical condensation technique. All treatments will be completed in a single session with the upper restorations. Patients will be given the VAS Pain Assessment Scale and asked to mark their individual pain levels between 0 and 10 at 6, 24, 48, 72 hours and 7 days after root canal treatment. At the end of the 7th day, patients will be called for a check-up and VAS questionnaires will be collected. Data will be collected in an excel table and analyzed.

Sample Size Calculation Sample size was calculated using the G*Power V. 3.1.9.6 program. Considering the pain values in the literature, it was decided to plan the study with a total of 60 cases, 20 in each group, with 95% confidence (1-α), 95% test power (1-β), f=0.412 effect size.* Considering the possible case losses as 20%, the final number of cases for each group will be 24.

Statistically Analysis Statistical analyses will be performed using the IBM SPSS Statistics for Windows, Version 25.0. (IBM Corp. Released 2017, Armonk, USA) package program. The package program has a license. Descriptive statistics will be given with percentage, frequency, mean ± standard deviation. Gender and age distributions according to groups were evaluated with Chi Square Analysis. Kruskal Wallis H test or ANOVA will be used to compare postoperative pain and according to VAS scores between three groups. Friedman Two-Way Variance Analysis will be used to evaluate VAS scores at all time points for each group. In case of significance, Dunn Test will be used by applying Bonferroni Correction in pairwise comparison of time points within groups. Significance level will be taken as α= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Patients who agreed to participate in this study
* Patients with single-canal, single-rooted teeth diagnosed with asymptomatic irreversible pulpitis due to trauma or deep carious lesions and patients with single-canal, single-rooted teeth referred for endodontic treatment for prosthetic reasons
* Patients with asymptomatic teeth
* Patients who have not used any analgesic, anti-inflammatory, or antibiotic drugs in the last 7 days
* Patients with good oral hygiene
* Patients with a sustained positive response to cold test and electric pulp test
* Patients with healthy periapical tissues (to be confirmed by periapical radiography)

Exclusion Criteria:

* Patients who refused to participate in this study
* Patients with medical problems (patients with immunosuppressive/systemic diseases, patients on medication)
* Patients with negative responses to thermal and electrical pulp tests
* Patients with advanced periodontal disease (probing depth >4 mm)
* Patients with preoperative percussion and palpation of the involved tooth
* Open apex, presence of calcification, presence of resorption
* Patients requiring endodontic treatment of more than one tooth
* Patients with allergic sensitivity to materials and agents to be used during root canal treatment
* Patients with allergic sensitivity to local anesthetics
* Patients with systemic or allergic sensitivity to NSAIDs
* Pregnant and lactating patients
* Teeth that cannot be restored due to excessive material loss in the coronal structure
* Overenstrumentation (extension of gutta-percha or root canal sealer beyond the radiographic apex) or short filling (more than 2 mm below the radiographic apex )
* Patients who develop acute exacerbations after the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 6th hour, 24th hour, 48th hour, 72nd hour, 7th day
  It is a system in which the patient marks the level of pain on a straight line divided from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yeniceri Ozata, Assoc Prof, Study Director — Dicle University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Dicle University, Faculty of Dentistry, Department of Endodontics, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will not share participants' personal data with third parties on this subject because I do not think it is right.

REFERENCES:
- [Result] Cosar M, Kandemir Demirci G, Caliskan MK. The effect of two different root canal sealers on treatment outcome and post-obturation pain in single-visit root canal treatment: A prospective randomized clinical trial. Int Endod J. 2023 Mar;56(3):318-330. doi: 10.1111/iej.13870. Epub 2022 Nov 22. PMID 36385378
- [Result] Ferreira NS, Gollo EKF, Boscato N, Arias A, Silva EJNLD. Postoperative pain after root canal filling with different endodontic sealers: a randomized clinical trial. Braz Oral Res. 2020;34:e069. doi: 10.1590/1807-3107bor-2020.vol34.0069. Epub 2020 Jul 15. PMID 32696911
- See also: Root canal obturation — https://endodontics.styleitaliano.org/root-canal-filling-systems-warm-vertical-condensation/